CLINICAL TRIAL: NCT03988387
Title: IPrEP, Study #2: Evaluating the Effectiveness, Feasibility and Acceptability of Enhanced Pre-exposure Prophylaxis (PrEP) Packages for Young Female Sex Workers in Kisumu, Kenya
Brief Title: IPREP Study #2: Evaluating Enhanced PrEP Packages for Young Female Sex Workers in Kisumu, Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Impact Research & Development Organization (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAS3722; R01MH110051 (NIH)
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: HIV
Keywords: Pre-exposure prophylaxis (PrEP); HIV prevention; Adherence
MeSH Terms: interventions — Emtricitabine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Peer Support PS) (Experimental): Participants randomized to the PS arm will be assigned a trained peer supporter (PSr) to enhance adherence to PrEP.
  Interventions: Behavioral: Peer Support (PS); Drug: daily oral PrEP (emtricitabine 200 mg/tenofovir 300 mg) [FTC/TDF]
- Reminders and Resource Transfer (RRT) (Experimental): Participants randomized to the RRT arm will receive weekly SMS text messages and resource transfers to enhance adherence to PrEP.
  Interventions: Behavioral: Reminder and Resource Transfer (RRT); Drug: daily oral PrEP (emtricitabine 200 mg/tenofovir 300 mg) [FTC/TDF]

INTERVENTIONS:
Behavioral: Peer Support (PS) — Participants randomized to the PS arm will be assigned a trained peer supporter. The peer supporters (PSr) will establish rapport and build trusting relationships with participants in order to increase self-efficacy and motivation to adhere to the daily PrEP regimen and to engage in HIV prevention behaviors, in general. The PSrs will assess for facilitators and barriers to PrEP adherence, conduct adherence counseling, and provide ongoing social and practical support (e.g. tailored appointment reminders, accompanying participants to medical appointments, and providing skills building for effective relationships with study site providers). PSrs will communicate with the participant on at least a weekly basis either in person or by phone and will track those who miss scheduled study visits. Participants will be encouraged to contact their PSrs in case of questions or concerns. For any clinical question, the peer supporter will direct the participant to the study nurse.
  Arms: Peer Support PS)
Behavioral: Reminder and Resource Transfer (RRT) — Participants who are randomized to the RRT arm will receive a discrete weekly SMS text (or voice message if participant is illiterate) to encourage healthy behaviors, study engagement and PrEP adherence. Messages will be a general message that the participant has selected and will not have any information identifying the participant as part of the study or describing the purpose of the study. An example text is "Remember to look after yourself today, See you tomorrow." Participants will be requested to respond to the message with a brief answer. Participants will be advised that each answered text counts as a point toward resource transfer that can be redeemed at scheduled study visits in the form of a small gift, such as cosmetics, personal care items, accessories, or airtime.The value of the reward increases with points.
  Arms: Reminders and Resource Transfer (RRT)
Drug: daily oral PrEP (emtricitabine 200 mg/tenofovir 300 mg) [FTC/TDF] — All participants will receive a one-month supply of daily oral PrEP (emtricitabine 200 mg/tenofovir 300 mg) [FTC/TDF] for the first month of enrollment.

SUMMARY:
This is an open-label randomized controlled trial (n=200) in which HIV-negative young female sex workers (FSW) will be randomized to receive oral PrEP combined with specific behavioral and structural adherence interventions, either: (1) Intensive Peer Support (PS) or (2) Reminders and Resource Transfer (RRT).Respondent-driven sampling (RDS) will be used to recruit FSW as potential study participants.The study adherence interventions will be delivered over the first 12-month period in conjunction with PrEP. Thereafter, the study-specific adherence interventions will be withdrawn and PrEP continued for an additional 12 months with standard support as per national guidelines. Trial participants will be followed for a total of 24 months and attend 11 study visits over this period.

DETAILED DESCRIPTION:
The overall aim of the proposed study is to compare the effectiveness, feasibility and acceptability of two adherence support interventions, peer support (PS) and reminders plus resource transfer (RRT), in combination with daily oral pre-exposure prophylaxis (PrEP) to optimize PrEP adherence among young in Kisumu, Kenya. Pre-exposure prophylaxis (PrEP) is a promising biomedical HIV prevention intervention. Findings from placebo-controlled efficacy trials highlight the need for adherence support to achieve PrEP efficacy and public health impact.

ELIGIBILITY:
Inclusion Criteria:

* Report no previous diagnosis of HIV infection
* Report being a cisgender female or transgender female
* Report being between 18-24 years of age
* Report living or working in study area
* Report intention to stay in study area for 24 months
* Report exchange sex with men for goods, money, favors or other services in past 3 months
* Report no previous or recent (within the last 3 months) PrEP use
* Able to complete study procedures in English, Kiswahili or Dholuo
* Willingness to be randomized and adhere to study interventions according to eligibility, including PrEP

Exclusion Criteria:

* Ineligible for PrEP according to Guidelines on Use of Antiretroviral Drugs for Treating and Preventing HIV Infection in Kenya - 2018 Edition (National AIDS and STI Control Program, 2018)
* Unable to provide informed consent for study procedures
* Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the principle investigators, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
* Reports plan to leave area in the next 24 months

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
PrEP Adherence between PS and RRT arms | 12 months
  Proportion of participants with ARV in plasma at 12-month visit

SECONDARY OUTCOMES:
PrEP Adherence between PS and RRT arms, any visit | At all visits
  Proportion of participants with detectable ARV in plasma at any visit
PrEP Adherence between PS and RRT arms, self-report | At all visits
  Proportion who report > 90% adherence by self-report
PrEP adherence across PS and RRT arms | 18 and 24 months
  Proportion of participants with ARV in plasma at 18- and 24- month visits
HIV risk behavior during PrEP use, propensity score | Baseline, 6, 12, 18, and 24 months
  Comparison of sexual risk propensity score
HIV risk behavior during PrEP use, unprotected sex | Baseline, 6, 12, 18, and 24 months
  Proportions of participants reporting unprotected vaginal or anal sex in the prior 30 days
Feasibility of PS and RRT interventions, intervention delivery | 24 months
  Proportion of expected intervention sessions delivered
Feasibility of PS and RRT interventions, study visit retention | 24 months
  Proportion of participants retained at each study visit
Completion of study visits between PS and RRT | 12, 18 and 24 months
  Proportion who completed scheduled PrEP study visits in PS and RRT arms at 18 and 24 months compared to proportion who completed these study visits at 12 months
Scaled perception of PrEP, PS and RRT | 24 months
  Scaled perceptions of satisfaction with and utility of PS and RRT intervention components, PrEP, and clinical care
Safety of PrEP including social harms | 24 months
  Discontinuation rates of PrEP due to an AE or drug toxicity and occurrence of social harms
Discontinuation of PrEP | 24 months
  Discontinuation rates of PrEP due to situational changes, dislike of PrEP

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa El-Sadr, MD, MPH, MPA, Principal Investigator — Columbia University
Locations (1):
- Tuungane Centre, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT03988387/ICF_000.pdf